CLINICAL TRIAL: NCT06660732
Title: A RandomizEd PhAse II TrIal of Rilonacept in Subjects With Cardiac Sarcoidosis (REPAIR-CS)
Brief Title: Rilonacept in Subjects With Cardiac Sarcoidosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Andrew N Rosenbaum, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-013175
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Cardiac Sarcoidosis
Keywords: Cardiac Sarcoidosis; Sarcoid Myocarditis; Myocarditis; Inflammation; PET scan; Heart Failure
MeSH Terms: conditions — Myocarditis; Inflammation; Heart Failure | interventions — rilonacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rilonacept+Standard therapy (Experimental)
  Interventions: Drug: Rilonacept
- Standard therapy (No Intervention)

INTERVENTIONS:
Drug: Rilonacept — 320 mg subcutaneous (SC) loading dose delivered as two 2-mL, subcutaneous injections of 160 mg on the same day at different anatomical sites followed by once weekly 160 mg SC doses.
  Other Names: KPL-914
  Arms: Rilonacept+Standard therapy

SUMMARY:
The primary objective of this study is to evaluate the effect of rilonacept, added to standard therapy and compared with standard therapy alone, on improvement in myocardial inflammation in subjects with cardiac sarcoidosis after 24 weeks of therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Able to comprehend and willing to sign an ICF and to abide by the study restrictions and requirements
2. Age ≥ 18 years and ≤ 80 years
3. Female subjects must be:

   * postmenopausal, defined as at least 12 months post cessation of menses (without an alternative medical cause), or
   * permanently sterile following documented hysterectomy, bilateral salpingectomy, bilateral oophorectomy, or tubal ligation, or having a male partner with vasectomy as affirmed by the subject, or
   * nonpregnant, nonlactating, and having agreed to use an effective method of contraception (i.e., hormonal contraception, intrauterine device [IUD], or double barrier methods such as condom plus diaphragm or diaphragm plus spermicide or condom plus spermicide) from Screening Visit 1 until 5 months after study drug administration, if sexually active.
4. Male subjects must have documented vasectomy or must use double barrier methods of contraception (such as condom plus diaphragm or diaphragm plus spermicide or condom plus spermicide) or use condoms plus hormonal contraceptives or condoms plus IUD with their female partners of childbearing potential from randomization to 3 months after the last dose of study drug administration. Male subjects must agree to refrain from donating sperm during this time period.
5. Routine adult vaccinations should be up to date and/or offered at least 2 weeks prior to randomization according to regional and national guidelines based on medical history or presence of risk factors, in the opinion of the Investigator.

   Cardiac Inclusion Criteria:
6. Has a diagnosis of cardiac sarcoidosis by the Heart Rhythm Society (HRS) expert consensus statement on the diagnosis and management of arrhythmias associated with cardiac sarcoidosis, or the Japanese Circulation Society 2016 Guideline on diagnosis and treatment of cardiac sarcoidosis (Terasaki 2019)
7. Three or more segments of active FDG uptake on PET scan within 8 weeks of randomization, despite standard therapy
8. Willing to wear an ambulatory cardiac rhythm monitor at the specified timepoints

Exclusion Criteria

1. Unable or unwilling to provide informed consent
2. Weight >380 pounds (172 kilograms)
3. Women who are pregnant or lactating or women of childbearing age who refuse to use a highly effective and medically acceptable form of contraception throughout the study
4. Planned to initiate TNF-α antagonist therapy over the course of the study.
5. Known claustrophobia, or difficulty completing prior PET scan procedure(s)
6. Left ventricular end-systolic diameter (LVESD) > 60 mm on echocardiogram
7. Other systemic immune disorder(s) or other disorder(s) that require treatment with immunomodulators or immunosuppressants
8. Has received, or is scheduled to receive after randomization, mechanical circulatory support
9. Congenital, valvular, and/or coronary artery disease that could explain the severity of cardiac dysfunction
10. Known hypersensitivity to rilonacept (KPL-914) or to any of its excipients
11. Meets the following TB criteria:

    1. History of active TB prior to screening OR
    2. History of latent TB that was not adequately treated prior to screening OR
    3. Signs or symptoms suggestive of active TB (e.g., new cough of >14 days in duration or a change in chronic cough, persistent fever, unintentional weight loss, or night sweats) upon review of medical history and/or physical examination at screening OR
    4. Recent close contact with a person with active TB OR
    5. Positive or indeterminate Interferon Gamma Release Assay (IGRA) test results or results from another positive TB test at screening based on acceptable local clinical practice
12. Use of the following immunosuppressive or immunomodulatory therapies (see also Section 5.6 "Prior and Concomitant Therapy") within the timeframe prior to randomization as defined below for each drug class or category:

    1. INCREASE in dose of existing immunosuppression/immunomodulation drug or INITIATION of new immunosuppression/immunomodulation drug in the one month prior to or ON or AFTER the date of the eligibility/baseline FDG-PET scan until the date of randomization.
    2. Anakinra within 1 week prior to first dose of study drug; canakinumab within 8 weeks prior to the first dose of study drug; abatacept within 8 weeks prior to first dose of study drug;
    3. TNF inhibitors within 2-8 weeks of or 5 half-lives (etanercept within 2 weeks; infliximab, certolizumab, golimumab, or adalimumab within 8 weeks) prior to first dose of study drug, whichever is longer.
    4. Rituximab within 6 months prior to the first dose of study drug unless levels of CD20+ B cells have been assessed and have returned to normal.
    5. Cyclosporine A (CsA) within 4 weeks prior to the first dose of study drug.
13. Received any investigational product within 30 days or 5 half-lives (if the half-life is known) of an investigational product (whichever is longer) prior to first dose of study drug
14. Concurrent enrollment in another clinical study, with the exception of observational studies
15. Uncontrolled hypertension (systolic blood pressure >170 mmHg and diastolic blood pressure >110 mmHg
16. Uncontrolled thyroid disease (serum TSH < 0.1 mU/L or > 10 mU/L)
17. Uncontrolled diabetes mellitus (serum glucose > 180 mg/dL fasting or HbA1c >9%)
18. Estimated glomerular filtration rate (eGFR) <30mL/min
19. Major surgery within 8 weeks prior to screening or planned major surgery within 6 months after first dose of study drug.
20. Transplanted organs (except corneal transplant performed more than 3 months prior to first dose of study drug).
21. Severe active, recurrent, or chronic infection (per PI discretion), or any episode of infection requiring hospitalization or treatment with a course of IV antibiotics within 12 weeks before screening. Subjects with a history of severe opportunistic infection (per PI discretion) are also excluded from the study.
22. High risk of infection (e.g., history of hereditary or acquired immune deficiency disorder), a history of an infected joint prosthesis at any time with that prosthesis still in situ, leg ulcers, indwelling urinary catheter, or persistent or recurrent chest infections.
23. Chronic active HBV infection, defined as:

    1. HBV surface antigen positive
    2. HBV anti-core antibody positive but anti-surface antibody negative
24. Presence of symptoms indicative of COVID-19 infection (per PI discretion), unless a PCR test for COVID-19 has been reported as negative within the previous 7 days or is acquired prior to randomization.
25. History of cancer within the last 5 years from screening, except for basal and squamous cell carcinoma of the skin or in situ carcinoma of the cervix treated and considered cured.
26. Has screening laboratory test results meeting any of the following criteria:

    1. Hemoglobin level < 8.0 g/dL
    2. WBC count < 3.0 × 103/µL
    3. Neutrophil count <1.5 × 103/µL
    4. Platelet count < 100 × 103/µL
    5. Total bilirubin level >1.5 × ULN unless the test results are consistent with those for Gilbert's syndrome
    6. AST or ALT values > 2 × ULN
27. Any condition that, in the opinion of the investigator, could interfere with evaluation of the investigational product or interpretation of subject safety or confound the results of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in number of segments with fluorodeoxyglucose F18 (FDG) uptake on cardiac fluorodeoxyglucose F18 - positron emission tomography (FDG-PET) scan | Baseline, Week 12, Week 24
  Fluorodeoxyglucose F18 uptake is evaluated across a 17 segment heart model. A higher number indicates higher myocardial inflammatory activity, while a lower number indicates lower inflammatory activity

SECONDARY OUTCOMES:
Change in maximum standardized uptake value (SUVMax) of the myocardium compared to baseline | Baseline, Week 12, Week 24
  Maximum standardized uptake is a ratio with the tracer uptake in region of interest / (injected activity / patient weight).
Summed perfusion rest score (SPRS) on fluorodeoxyglucose F18 - positron emission tomography (FDG-PET) scan | Week 24
  Summed perfusion rest score (SPRS) provides an overall assessment of myocardial perfusion. A higher score reflects worse perfusion, and a lower score reflects better perfusion.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Rosenbaum, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No